CLINICAL TRIAL: NCT05458492
Title: Cutaneous Sarcoidosis With Moderate to Severe Involvement of the Face : Multicenter Open-label Study of Oral Sirolimus Efficacy and Tolerance
Brief Title: Sirolimus in Cutaneous Sarcoidosis
Acronym: SIRIUS
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APHP180156
Record Dates: First submitted 2021-10-11; First posted 2022-07-14 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: Sarcoidosis; Cutaneous Sarcoidosis
MeSH Terms: conditions — Sarcoidosis | interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sirolimus Arm (Experimental): Sirolimus, tablets 2 mg/day with dose adjustment of 1 to 3 mg/day for residual concentrations between 4 and 10 ng/mL
  1 dose daily for 16 weeks
  Interventions: Drug: Sirolimus

INTERVENTIONS:
Drug: Sirolimus — Sirolimus, tablets 2 mg/day with dose adjustment of 1 to 3 mg/day for residual concentrations between 4 and 10 ng/mL
  1 dose daily for 16 weeks

SUMMARY:
Sarcoidosis is a multisystemic disease of unknown etiology characterized by the presence of epithelioid granulomas without caseous necrosis in the organs involved. Sarcoidosis cutaneous lesions can be severe. There is no recommendation for the treatment of cutaneous sarcoidosis. A recent study highlights the potential efficacy of mTOR inhibitors in the treatment of sarcoidosis granulomas. The hypothesis is that sirolimus could be effective for sarcoidosis treatment, especially for cutaneous lesions.

The main objective of this study is to evaluate sirolimus efficacy on cutaneous sarcoidosis of the face.

The main evaluation criteria is the percentage of patients with a significant clinical response (relative decrease in "facial SASI" ≥ 25%) at week 16 of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old <75 years old (men and women)
* Cutaneous sarcoidosis of the face (diagnosed according to the following criteria : compatible clinical appearance showing erythemato-purple, brownish or yellowish macules or papules or nodules and compatible histological appearance with a facial or extra facial skin biopsy confirming the diagnosis of sarcoidosis showing epithelioid and giganto-cellular granuloma without caseous necrosis) moderate to severe defined by: "Facial SASI" Score (Sarcoidosis Area and Severity Index) ≥ 2 and PGA (Physician's Global Assessment,0 to 10 scale) ≥ 5
* Health insurance plan coverage
* Patients who never had a systemic treatment or who had at least one classical systemic treatment failure for sarcoidosis treatment
* For women of childbearing age (unless post-menopausal or sterile), pregnancy test with βHCG negative. Effective contraception should be used during sirolimus treatment and for 12 weeks after stopping sirolimus
* Patients who have signed a written consent

Exclusion Criteria:

* Severe hepatic failure (Cytolysis (ALAT)> 3N and / or Cholestase (PAL)> 3N)
* Allergy or intolerance to sirolimus or at one of its excipients
* Allergy to peanut or soybeans
* Patient with a pulmonary or hepatic graft
* General corticotherapy or immunosuppressive treatment (methotrexate, azathioprine, mycophenolate mofetil, cyclophosphamide, ciclosporin) in the month before the inclusion
* Intra-lesional corticotherapy for less than 3 months
* Biotherapy (anti-TNFa, anti-IL12/23, anti-IL17A) within 3 months preceding the inclusion
* Thalidomide or other -imide treatment for less than 3 months
* Cyclins treatment for less than 1 month
* Topical corticosteroids or topical tacrolimus for less than 1 week
* Sarcoidosis involvement of at least one organ requiring systemic treatment other than sirolimus (oral corticosteroid or systemic immunosuppressive treatment)
* Cholesterolemia> 300 mg/ dl or triglyceridemia> 400 mg/dl
* Administration of strong CYP3A4 inhibitors or inducers such as rifampicin, ketoconazole, voriconazole, telithromycin , diltiazem, verapamil, erythromycin, clarythromycin, ciclosporin
* Pregnancy or breastfeeding
* Active infection including tuberculosis disease
* Non-controlled arterial hypertension (TAS> 150 mmHg and / or TAD> 100 mmHg)
* Patient under guardianship or curatorship, patients deprived of freedom, under safeguarding of justice, receiving psychiatric care, under the constraint, admitted in a health or social institution for purposes other than those of research
* Patient with cancer (except cutaneous basal cell carcinoma or in situ cervical cancer)
* Risk of patient bad compliance
* Grapefruit or grapefruit juice consumption during the treatment duration
* Patients with fructose intolerance, galactose intolerance, glucose-galactose malabsorption, insufficiency in sucrase-isomaltase or Lapp lactase

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-07 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with a significant clinical response | at week 16
  Significant clinical response will be defined as a relative decrease in "facial SASI" ≥ 25% compared to baseline.
  Facial SASI score evaluates 4 features for each of 4 facial quadrants and the nose: erythema, induration, and desquamation, each ranging from 0 (none) to 4 (very severe), and an area score ranging from 0 (0%) to 6 (90-100%). The maximal range of modified Facial SASI scores is 0 to 72.

SECONDARY OUTCOMES:
Percentage of patients with a good clinical response | at week 16
  A good clinical response will be defined as a relative decrease of "facial SASI" ≥ 50%.
  Facial SASI score evaluates 4 features for each of 4 facial quadrants and the nose: erythema, induration, and desquamation, each ranging from 0 (none) to 4 (very severe), and an area score ranging from 0 (0%) to 6 (90-100%). The maximal range of modified Facial SASI scores is 0 to 72.
Percentage of patients with complete clinical response | at week 16
  Complete clinical response will be defined as "facial SASI" = 0. Facial SASI score evaluates 4 features for each of 4 facial quadrants and the nose: erythema, induration, and desquamation, each ranging from 0 (none) to 4 (very severe), and an area score ranging from 0 (0%) to 6 (90-100%). The maximal range of modified Facial SASI scores is 0 to 72.
Percentage of patients with an improvement of their quality of dermatological life | at week 16
  An improvement will be defined as a decrease of Dermatology Life Quality Index (DLQI) questionnaire> 25%. DLQI goes from 0 to 30. A lower score indicated a good quality of Life, and a higher score a worse quality of life.
Comparison of face facial photographs with good brightness compared to baseline | at week 16
  Qualitative clinical aspects of skin sarcoidosis lesions will be compared between baseline and Week 16, as an illustrative proof in addition to quantitative skin score assessment (Facial SASI)
Sarcoidosis activity score evaluated for other organs evaluted using Extra-Pulmonary Physician Organ Severity Tool (ePOST) | at week 16
  Sarcoidosis activity for all organs will be evaluted using Extra-Pulmonary Physician Organ Severity Tool (ePOST) (from 0 (normal) to 6(severe impairment))
Sarcoidosis activity score evaluated for other organs evaluted using Extra-Pulmonary Physician Organ Severity Tool (ePOST) | at 12 months
  Sarcoidosis activity for all organs will be evaluted using Extra-Pulmonary Physician Organ Severity Tool (ePOST) (from 0 (normal) to 6(severe impairment))
Sarcoidosis activity score evaluated for other organs using Score Sarcoidosis disease activity index (SDAI score) | at 16 weeks
  Sarcoidosis activity for all organs will be evaluted using Score Sarcoidosis disease activity index (SDAI score) : it goes from 0 to 167 (the higher the score, the greater the disease activity).
Sarcoidosis activity score evaluated for other organs using Score Sarcoidosis disease activity index (SDAI score) | at 12 months
  Sarcoidosis activity for all organs will be evaluted using Score Sarcoidosis disease activity index (SDAI score) : it goes from 0 to 167 (the higher the score, the greater the disease activity).
Pulmonary Sarcoidosis activity | at week 16
  Pulmonary Sarcoidosis activity will be assessed using Abbreviated CT score to quantify disease activity in pulmonary sarcoidosis (aCTAS score) to assess pulmonary involvement. It goes from 0 to 4 (the higher the score, the greater the pulmonary disease activity).
Pulmonary Sarcoidosis activity | at 12 months
  Pulmonary Sarcoidosis activity will be assessed using Abbreviated CT score to quantify disease activity in pulmonary sarcoidosis (aCTAS score) to assess pulmonary involvement. It goes from 0 to 4 (the higher the score, the greater the pulmonary disease activity).
Pulmonary sarcoidosis functionnal evaluation assessed using Functional respiratory explorations by vital capacity | at week 16
  Pulmonary sarcoidosis functionnal evaluation will be assessed using Functional respiratory explorations by vital capacity
Pulmonary sarcoidosis functionnal evaluation assessed using Functional respiratory explorations by vital capacity | at 12 months
  Pulmonary sarcoidosis functionnal evaluation will be assessed using Functional respiratory explorations by vital capacity
Pulmonary sarcoidosis functionnal evaluation assessed by walking perimeter | at week 16
  Pulmonary sarcoidosis functionnal evaluation will be assessed by walking perimeter (in meters)
Pulmonary sarcoidosis functionnal evaluation assessed by walking perimeter | at 12 months
  Pulmonary sarcoidosis functionnal evaluation will be assessed by walking perimeter (in meters)
Percentage of patients with adverse events | up to 16 weeks
Evaluate CD68, phospho-mTOR and phospho-p70S6K expression on skin biopsies | at 16 weeks
  Immunohistochemical assessment will be assessed using optical microscopy
Transcriptomic analysis of skin | at 16 weeks
  It will be assessed using microarray (Affymetrix)
Circulating monocytes | at 16 weeks
  It will be assessed using microarray (Affymetrix)
Percentage of patients with a complete or near-complete response based on PGA (PGA = 0 or 1) of the skin. | at 16 weeks

IPD SHARING:
Plan to Share IPD: Undecided